CLINICAL TRIAL: NCT00093418
Title: Phase II Studies of Two Different Schedules and Two Different Doses of the Farnesyl Transferase Inhibitor R115777 (Tipifarnib, Zarnestra®, NSC-702818) for Previously Untreated Acute Myeloid Leukemia (AML) in Patients of Age 70 or Older
Brief Title: S0432 Tipifarnib in Treating Older Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03038; S0432; U10CA032102 (NIH); CDR0000387957 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — tipifarnib

ARMS (4):
- Arm I (Experimental): Arm I: Patients receive oral tipifarnib twice daily on days 1-21. In all arms, courses repeat every 28 days in the absence of unacceptable toxicity or disease progression. Patients who achieve a complete remission (CR) receive up to 3 additional courses beyond CR. Patients in CR who develop recurrent disease after the completion of therapy are eligible to receive tipifarnib again.
  Interventions: Drug: tipifarnib
- Arm II (Experimental): Patients receive oral tipifarnib twice daily on days 1-7 and 15-21. In all arms, courses repeat every 28 days in the absence of unacceptable toxicity or disease progression. Patients who achieve a complete remission (CR) receive up to 3 additional courses beyond CR. Patients in CR who develop recurrent disease after the completion of therapy are eligible to receive tipifarnib again.
  Interventions: Drug: tipifarnib
- Arm III (Experimental): Patients receive tipifarnib as in arm I, but at a lower dose. In all arms, courses repeat every 28 days in the absence of unacceptable toxicity or disease progression. Patients who achieve a complete remission (CR) receive up to 3 additional courses beyond CR. Patients in CR who develop recurrent disease after the completion of therapy are eligible to receive tipifarnib again.
  Interventions: Drug: tipifarnib
- Arm IV (Experimental): Patients receive tipifarnib as in arm II, but at a lower dose. In all arms, courses repeat every 28 days in the absence of unacceptable toxicity or disease progression. Patients who achieve a complete remission (CR) receive up to 3 additional courses beyond CR. Patients in CR who develop recurrent disease after the completion of therapy are eligible to receive tipifarnib again.
  Interventions: Drug: tipifarnib

INTERVENTIONS:
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra

SUMMARY:
This randomized phase II trial is studying 4 different tipifarnib regimens to compare how well they work in treating older patients with acute myeloid leukemia. Tipifarnib may stop the growth of cancer cells by blocking the enzymes necessary for their growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test whether any or all of four different regimens of R115777 (tipifarnib) is sufficiently effective therapy for previously untreated acute myeloid leukemia (AML) in patients of age 70 or older to warrant Phase III investigation. Additionally, to allow increased access for patients to an agent that appears promising in this patient population.

II. To estimate the frequency and severity of toxicities of these regimens in this group of patients.

III. To investigate in a preliminary manner the relationship of cytogenetics with response to R115777 (tipifarnib) and assess whether karyotype represents a potential prognostic factor among older AML patients who are not candidates for chemotherapy and are treated with R1157777.

IV. To collect specimens for future correlations (e.g. RAS and downstream targets) to be identified at a later date.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 4 treatment arms.

ARM I: Patients receive oral tipifarnib twice daily on days 1-21. ARM II: Patients receive oral tipifarnib twice daily on days 1-7 and 15-21. ARM III: Patients receive tipifarnib as in arm I, but at a lower dose. ARM IV: Patients receive tipifarnib as in arm II, but at a lower dose.

In all arms, courses repeat every 28 days in the absence of unacceptable toxicity or disease progression. Patients who achieve a complete remission (CR) receive up to 3 additional courses beyond CR. Patients in CR who develop recurrent disease after the completion of therapy are eligible to receive tipifarnib again.

Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a morphologically confirmed diagnosis of acute myeloid leukemia (AML) with classification other than WHO Acute Promyelocytic Leukemia (FAB M3), based on bone marrow aspiration and biopsy performed within 14 days prior to registration; if a diagnostic biopsy has been performed within 28 days prior to registration, the marrow blast percentage is >= 70%, and no potentially anti-leukemic therapy has been given in the interim, then this bone marrow examination can be used for registration purposes; Note: This protocol uses the WHO diagnostic criteria for AML, not the FAB criteria; patients with WHO Acute Promyelocytic Leukemia (FAB M3) or blastic transformation of chronic myelogenous leukemia are not eligible; patients must not be candidates for or must have refused standard AML cytotoxic chemotherapy regimens
* Patients must not have received prior systemic chemotherapy for acute leukemia with the exception of hydroxyurea; patients must have a WBC =< 30,000/cmm within 1 day prior to registration; administration of hydroxyurea to control high WBC count prior to, during and after registration is permitted; patients with a history of prior myelodysplastic syndrome are eligible; however, prior treatment with AML induction type chemotherapy or high dose chemotherapy with hematopoietic stem cell support is not allowed; patients may have received hematopoietic growth factors, thalidomide, arsenic trioxide, signal transduction inhibitors, azacitidine, and low dose cytarabine for treatment of myelodysplastic syndrome; however, the dose of cytarabine must be < 100 mg/M2/day; other low intensity therapies for MDS will also be permitted and should be discussed with the Study Coordinator; patients must be off prior therapy for MDS (excluding growth factors) and all toxicities must have resolved; if indicated, a single dose of intrathecal chemotherapy may also be given before or concurrent with induction chemotherapy
* Patient must have a bilirubin =< 1.5 x Institutional Upper Limit of Normal (IULN), unless the elevation is due primarily to elevated unconjugated hyperbilirubinemia secondary to Gilbert's syndrome or hemolysis and not to liver dysfunction
* SGOT (AST) =< 2.5 x IULN, or SGPT (ALT) =< 2.5 x IULN, or both within 14 days prior to registration
* Patients must have a serum creatinine =< 1.5 x IULN within 14 days prior to registration
* Southwest Oncology Group patients must be registered on SWOG-9007, the cytogenetics protocol; collection of pretreatment marrow specimens must be completed within 14 days prior to registration; pretreatment specimens of bone marrow must be submitted to an approved Southwest Oncology Group Cytogenetics Laboratory for cytogenetic analysis; note that protocol SWOG-9007 also requires submission of remission and relapse specimens
* ECOG and CALGB have similar cytogenetics studies; please check with your group to find out about requirements for participation; CTSU sites will not be participating in SWOG-9007 and will not be submitting specimens for this study
* All patients must have cytogenetics performed and - if not registered to SWOG-9007 - a cytogenetics report submitted to the Cytogenetics Office at the Southwest Oncology Group Data Operations Center
* Southwest Oncology Group patients must be offered participation in S9910, the leukemia centralized reference laboratories and tissue repositories ancillary study; if consent is given, collection of pretreatment blood and/or marrow specimens must be completed within 14 days prior to registration; if the patient consents to participate in S9910, pretreatment specimens of marrow and/or peripheral blood must be submitted to the Southwest Oncology Group Myeloid Repository at the University of New Mexico for cellular and molecular studies; S9910 also requests submission of remission and relapse specimens
* ECOG and CALGB have similar reference laboratories and repository protocols; please check with your group to find out about requirements for participation
* CTSU sites will not be participating in S9910 and will not be submitting specimens for this study
* Patients of reproductive potential must have agreed to use an effective contraceptive method
* Patients with a prior malignancy are eligible; however, the patient must have completed all chemotherapy and radiotherapy at least 6 months prior to study registration; there should be no plan to begin therapy for the prior malignancy at the time of study registration; concurrent hormonal therapy is allowed
* Patients who are expected to require treatment with enzyme inducing antiepileptic drugs (EIAED) are not eligible for this study
* If day 14 or 30 falls on a weekend or holiday, the limit may be extended to the next working day; in calculating days of tests and measurements, the day a test or measurement is done is considered Day 0; therefore, if a test is done on a Monday, the Monday two weeks later would be considered Day 14; this allows for efficient patient scheduling without exceeding the guidelines
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 296 (Actual)
Dates: Start 2004-09; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Total response rate, defined as the proportion of patients who achieve CR or PR | Up to 3 years
  Any of the regimens considered in this trial would be considered sufficiently promising for further study if it increased the true total response rate of 30%, but not sufficiently promising if it produced a true total response rate of only 10%.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Erba, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States